CLINICAL TRIAL: NCT06262295
Title: France LEADLESS, a Safety and Effectiveness Monitoring in France for AVEIR VR LP and AVEIR AR LP
Brief Title: A Safety and Effectiveness Monitoring in France for AVEIR VR LP and AVEIR AR LP
Acronym: France LEADLES
Status: Recruiting | Type: Observational
Sponsor: French Cardiology Society (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A02475-40
Record Dates: First submitted 2024-02-06; First posted 2024-02-16 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Pacemaker
Keywords: Leadless stimulator; Pacemaker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subject is going to or has been implanted with an AVEIR VR LP device and/or an AR LP device

SUMMARY:
Although the idea of a leadless pacemaker was first proposed in the 1970s to eliminate the probes, pockets and connectors required by conventional cardiac procedures and the associated complications, the first devices were not developed until the late 2010s. Leadless pacemakers can also improve patient comfort by replacing surgery with a percutaneous procedure, eliminating the mass and scar visible at the implantation site of a conventional pacemaker, and eliminating the need for activity restrictions to prevent dislodgement after implantation of a conventional lead.

This french Registry "France LEADLESS" is a national registry designed to confirm the safety and efficacy of the AVEIR VR LP System in a patient population indicated for the implantation of a VVI(R) pacemaker in France and the AVEIR AR LP System in a population of patients indicated for the implantation of an AAI(R) pacemaker or both systems used in conjunction in a population of patients indicated for the implantation of a DDD(R) pacemaker. This registry will also make it possible to collect the characteristics and indications of patients under normal conditions of use.

DETAILED DESCRIPTION:
Observational national multicentric registry. Retrospective and Prospective, non-randomized, single-arm allowing exhaustive follow up of all AVEIR VR and AR LP implants in France.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with an AVEIR VR LP device and/or an AR LP device
* Patient over 18 years old
* Patient informed of the nature of the study, agrees to participate in the study

Exclusion Criteria:

* Patient under 18 years of age
* Patient refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included in cardiology departments participating in the study. This french Registry "France LEADLESS" is a national registry designed to confirm the safety and efficacy of the AVEIR VR LP System in a patient population indicated for the implantation of a VVI(R) pacemaker in France and the AVEIR AR LP System in a population of patients indicated for the implantation of an AAI(R) pacemaker or both systems used in conjunction in a population of patients indicated for the implantation of a DDD(R) pacemaker.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2028-09-14 (Estimated); Study Completion 2028-09-14 (Estimated)

PRIMARY OUTCOMES:
To confirm the safety of the AVEIR VR LP device and/or an AR LP device | during 24 months after implantation
  Assessed by rate of successful implantation, absence of complications (as assessed by number of procedural or device related complications) and reoperation (as assessed by number of replacement, explantation, change in device position)
To confirm the effectiveness of the AVEIR VR LP device and/or an AR LP device | during 24 months after implantation
  device longevity
To confirm the effectiveness of the AVEIR VR LP device and/or an AR LP device | during 24 months after implantation
  electrical performance of the device
To collect patient characteristics and indications in normal conditions of use of the AVEIR VR LP device and/or an AR LP device | during 24 months after implantation
  Exhaustive collection of all cases of patients implanted in all French centers accredited to implant leadless stimulators in France

CONTACTS AND LOCATIONS:
Overall Officials: Pascal DEFAYE, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- Chu de Grenoble - Hopital Michallon, La Tronche, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Eur Heart J. 2021 Sep 14;42(35):3427-3520. doi: 10.1093/eurheartj/ehab364. No abstract available. PMID 34455430
- [Background] Udo EO, Zuithoff NP, van Hemel NM, de Cock CC, Hendriks T, Doevendans PA, Moons KG. Incidence and predictors of short- and long-term complications in pacemaker therapy: the FOLLOWPACE study. Heart Rhythm. 2012 May;9(5):728-35. doi: 10.1016/j.hrthm.2011.12.014. Epub 2011 Dec 17. PMID 22182495
- [Background] Kirkfeldt RE, Johansen JB, Nohr EA, Jorgensen OD, Nielsen JC. Complications after cardiac implantable electronic device implantations: an analysis of a complete, nationwide cohort in Denmark. Eur Heart J. 2014 May;35(18):1186-94. doi: 10.1093/eurheartj/eht511. Epub 2013 Dec 17. PMID 24347317
- [Background] Reddy VY, Knops RE, Sperzel J, Miller MA, Petru J, Simon J, Sediva L, de Groot JR, Tjong FV, Jacobson P, Ostrosff A, Dukkipati SR, Koruth JS, Wilde AA, Kautzner J, Neuzil P. Permanent leadless cardiac pacing: results of the LEADLESS trial. Circulation. 2014 Apr 8;129(14):1466-71. doi: 10.1161/CIRCULATIONAHA.113.006987. Epub 2014 Mar 24. PMID 24664277
- [Background] Knops RE, Tjong FV, Neuzil P, Sperzel J, Miller MA, Petru J, Simon J, Sediva L, de Groot JR, Dukkipati SR, Koruth JS, Wilde AA, Kautzner J, Reddy VY. Chronic performance of a leadless cardiac pacemaker: 1-year follow-up of the LEADLESS trial. J Am Coll Cardiol. 2015 Apr 21;65(15):1497-504. doi: 10.1016/j.jacc.2015.02.022. PMID 25881930